CLINICAL TRIAL: NCT04056364
Title: Diagnostic Value of Sputum Cytology in Asthma-COPD Overlap
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Memo Ahmed, Principal Investigator, Assiut University
Other Study IDs: sputum cytology
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: COPD, Asthma,ACO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthma: Asthma patients will be diagnosed according to a clinical history of wheezing, cough, chest tightness or shortness of breath, as well as the presence of BHR (cumulative dose caus¬ing a 20% decrease in FEV1), based on the GINA guidelines. None of them had a history of COPD, or previous doctor-diagnosed ACO. All subjects had not used any oral or/and inhaled corticosteroid (ICS) in the previous 12 weeks. The included patients with asthma had initial diagnosis and were under uncontrolled stage.
  Interventions: Biological: sputum cytology
- COPD: COPD patients were diagnosed according to the GOLD criterion, which included a post-bronchodilator spirometry to confirm airflow obstruction (FEV1 to forced vital capacity ratio [FEV1/FVC] ,70%), in a clinical context (dyspnea, chronic cough or sputum production, and a history of expo¬sure to risk factors for the disease). They had received a COPD diagnosis at least 1 year before the study. None of them had a history of asthma. All subjects had not used any oral or/and ICS in the previous 4 weeks. The included COPD patients had exacerbations. The GOLD stage of COPD was defined according to the 2019 recommendations of GOLD.
  Interventions: Biological: sputum cytology
- ACO: ACO will be diagnosed by two steps: the first step is the identification of a history of chronic airway disease, i.e., chronic or recurrent cough, sputum production, wheezing, or repeated acute lower respiratory tract infections. In the second step, the features of asthma and those of COPD that best describe the patients
  Interventions: Biological: sputum cytology

INTERVENTIONS:
Biological: sputum cytology — Sputum cytology refers to the examination of sputum (mucus) under a microscope to look for abnormal or cancerous cells. Sputum, or phlegm, is the fluid that is secreted by cells in the lower respiratory tract such as the bronchi and the trachea. It differs from saliva, in that it contains cells that line the respiratory passages.

SUMMARY:
The aim of this study is to evaluate the diagnostic value of sputum cell counts in differentiation between asthma, COPD and ACO.

to examine the relationship between sputum cell counts in bronchial revers¬ibility and bronchial hyperresponsiveness

DETAILED DESCRIPTION:
Asthma and COPD are considered as chronic airway inflammatory diseases, which are typically associated with Th2-mediated immune response in asthma and related to the characteristics of Th1-mediated immunity in COPD . Asthma-COPD overlap (ACO) is the term to describe patients who have features of both asthma and COPD, recom¬mended by the 2019 Global Initiative for Asthma (GINA) and the Global Initiative for Chronic Obstruction Lung Disease (GOLD) guidelines. Patients with asthma and COPD are commonly seen in clinical practice. In addition, compared with patients with asthma or COPD alone, patients with ACO experience frequent exacerbations and hospitalizations, have poor quality of life, a more rapid decline in lung function and high mortality, and consume a disproportionate amount of health care resources than asthma or COPD alone .

Cell count in induced sputum is a noninvasive biomarker to assess airway inflammation phenotypes. Accordingly, sputum cell counts are extensively used in the treatment of asthma and COPD. Nevertheless, the clinical application of sputum cell counts in patients with asthma-COPD overlap (ACO) remains elusive .

ELIGIBILITY:
Inclusion Criteria:

* all patients known to be Asthma, COPD, ACO

Exclusion Criteria:

* Patients will be excluded if they have confounding pulmonary comorbidities, such as pulmonary tuberculosis, interstitial lung disease, lung cancer or pulmonary infection, and had a cognitive impairment that may affect the collaboration or comprehension of the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients known have Asthma, COPD, ACO . age from 18 years until 75
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
comparison of sputum cytology in Asthma , COPD, ACO | Baseline
  A differential cell count will be obtained from 400 cells under 400× microscope to identify the severity and type of airway inflammation in all patients. Squamous cell count less than 10% in each sample will be deemed adequate for further analysis.

REFERENCES:
- [Background] Ojanguren I, Moullec G, Hobeika J, Miravitlles M, Lemiere C. Clinical and inflammatory characteristics of Asthma-COPD overlap in workers with occupational asthma. PLoS One. 2018 Mar 2;13(3):e0193144. doi: 10.1371/journal.pone.0193144. eCollection 2018. PMID 29499062